CLINICAL TRIAL: NCT03892668
Title: Safety and Efficacy of Intravenous Oxytocin Versus Tranexamic Acid in Reducing Blood Loss During Abdominal Myomectomy; A Randomized Controlled Trial
Brief Title: Intravenous Oxytocin Versus Tranexamic Acid in Reducing Blood Loss During Abdominal Myomectomy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor of obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: myomectomy
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Myomectomy
MeSH Terms: interventions — Tranexamic Acid; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tranexamic acid (Experimental): Patients in the TXA group will be given 15 mg/kg of tranexamic acid (Cyklokapron@; Amoun Pharmaceutical Co., SAE) slowly intravenously 30 min before surgery followed by 10 mg/ kg/h infusion in 500 ml Ringer's by infusion pump till the end of the procedure.
  Interventions: Drug: Tranexamic Acid
- oxytocin (Active Comparator): An equal volume of normal saline syringe in a double blinded manner will be intravenously administered to the OXYtocin group 30 min before surgery and will be followed by one ampoule of oxytocin (10 U/mL/amp) (Syntocinon; Aventis Pharmaceutical Co.) will be added to 500 mL Ringer's solution running at a rate of 400 mU/min by infusion pump till the end of the procedure.
  Interventions: Drug: oxytocin
- placebo (Placebo Comparator): An equal volume of normal saline syringe in a double blinded manner will be intravenously administered to the oxytocin group 30 min before surgery and will be followed by 500 ml saline infusion during the operation
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Patients in the TXA group will be given 15 mg/kg of tranexamic acid (Cyklokapron@; Amoun Pharmaceutical Co., SAE) slowly intravenously 30 min before surgery followed by 10 mg/ kg/h infusion in 500 ml Ringer's by infusion pump till the end of the procedure.
  Arms: tranexamic acid
Drug: oxytocin — An equal volume of normal saline syringe in a double blinded manner will be intravenously administered to the OXYtocin group 30 min before surgery and will be followed by one ampoule of oxytocin (10 U/mL/amp) (Syntocinon; Aventis Pharmaceutical Co.) will be added to 500 mL Ringer's solution running at a rate of 400 mU/min by infusion pump till the end of the procedure.
  Arms: oxytocin
Drug: placebo — An equal volume of normal saline syringe in a double blinded manner will be intravenously administered to the Oxytocin group 30 min before surgery and will be followed by 500 ml saline infusion during the operation
  Arms: placebo

SUMMARY:
Uterine leiomyomas (fibroids) are the most common benign tumors among women. Fibroids are found in approximately 20% of women over 35 years of age. In 20-50% of patients, fibroids may cause problems such as heavy menstrual bleeding, anemia, pelvic pain, pressure symptoms from extrinsic compression of the colorectal and urinary tract. Surgery is indicated for symptomatic uterine leiomyomas; hysterectomy for women who have completed childbearing (women > 40 years old), and myomectomy for women <40 years old who wish to preserve uterus and fertility.

DETAILED DESCRIPTION:
Interventions:

Preoperative

* Full history, where demographic characteristics will be reported and examination to detect the size and mobility of uterus.
* Informed consent will be taken from patients.
* Trans-vaginal U/S to assess number, size, and types of myomas.
* Preoperative full labs (Hemoglobin, hematocrit, INR, liver enzymes and kidney functions)

Intra Operative

* Preoperative antibiotics will be given before the beginning of the operation. The operations will be performed as standard through a midline or Pfannenstiel incision by the same consultant gynecologist to ensure consistency of study procedures. All patients will receive general anesthesia. After the skin incision, the subcutaneous fat and abdominal fascia will be opened crosswise, and the rectus muscle will be opened on the midline. The parietal peritoneum will be opened longitudinally to reach the pelvic cavity. Subsequently, a self-retaining retractor will be inserted, and intestine will be packed. The uterus will be inspected for the number, location, and shape of myomas. Other pelvic organs will be inspected for any associated pathology. When possible, uterine incisions will be performed on the anterior wall or fundus in order to reduce postoperative adhesions. The incision will be performed using monopolar diathermy. Intracapsular enucleation of myomas will be performed by gently dissecting between the myoma and the pseudo-capsule. The myoma will be gently enucleated out. Meticulous hemostasis will be secured by low-voltage coagulation of feeding vessels. Myoma bed will be closed by 1 or 2 layers of interrupted vicryl sutures (Vicryl 1-0 polyglactin 910; Egycryl, Taisier CO, Egypt). No mechanical tourniquet or local vasoocclusive drugs (e.g., vasopressin) will be used intraoperatively.
* The study will include patients scheduled for open abdominal myomectomy and will be divided into three equal groups.
* All the three groups will take a standard dose of 400 microgram of misoprostol rectally one hour before the operation.

Postoperative

* Estimation of Hemoglobin 6 hrs postoperatively and next day morning.
* Monitor Vital Signs and need for blood transfusion.
* Send myomas for pathology.

ELIGIBILITY:
Inclusion Criteria:

* • Age group (18-50) years old

  * Intramural or interstitial myomas (more than 5 cm)
  * Symptomatic myomas (heavy menstrual bleeding or pain during menstruation)
  * Abdominal myomectomy
  * No medical disorders
  * No coagulation disorders

Exclusion Criteria:

* • Age group (less than 18 yrs old)

  * Age group (more than 50 yrs old)
  * Subserous or submucous myomas
  * Laparoscopic or hysteroscopic myomectomy
  * Medical disorders (for example uncontrolled hypertension, diabetes mellitus, renal or hepatic disorders)
  * Coagulation disorders
  * Previous use of anticoagulant drugs
  * Previous myomectomy
  * Allergy to Tranexamic acid or oxytocin
  * Malignant features by U/S or examination
  * Pregnancy
  * Previous hormonal therapy (GnRH analogues)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Intraoperative Blood loss | during the operation
  The total volume of intraoperative blood loss was estimated by measuring the amount of blood accumulated in the aspiration equipment and the amount of blood on the surgical gauze using an alkaline hematin technique

SECONDARY OUTCOMES:
Operation time | 1 hour
  Operation time from skin incision to skin closure in minutes.
Myomectomy time | 30 minutes
  Myomectomy time from first uterine incision to closure of last uterine incision in minutes

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine Cairo university, Giza, Egypt